CLINICAL TRIAL: NCT07110155
Title: Is the Evolution of the Aldosterone-renin Ratio Pre- Versus Post-operative on Day 1 Following Unilateral Adrenalectomy for Primary Hyperaldosteronism Predictive of Blood Pressure Outcomes
Acronym: vRAR
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, NOMINE-CRIQUI Claire, PH, Central Hospital, Nancy, France
Other Study IDs: 2025PI029
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Hyperaldosteronism Primary
Keywords: arterial hypertension; unilateral adrenalectomy; aldosterone-to-renin ratio (ARR)
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent unilateral adrenalectomy for primary hyperaldosteronism between 2017 and 2025

SUMMARY:
Primary hyperaldosteronism is characterised by excessive and autonomous aldosterone secretion by the adrenal glands, independent of renin. The condition is characterised by an aldosterone-to-renin ratio (ARR) that exceeds a certain pathological threshold. It manifests as arterial hypertension, which is potentially associated with hypokalaemia due to increased urinary potassium excretion. Excessive and unregulated aldosterone secretion is a validated risk factor for cardiovascular complications.

Primary hyperaldosteronism is estimated to account for 5-20% of hypertension cases and up to 25% of resistant hypertension cases.

Autonomous aldosterone secretion may originate from unilateral secretion by a benign adrenal cortical tumour (Conn's adenoma). Treatment usually involves surgical removal of the hypersecretion source via unilateral adrenalectomy. Alternatively, it can correspond to bilateral adrenal secretion, with or without lateralisation (bilateral adrenal hyperplasia), which is typically managed with antihypertensive medications and/or mineralocorticoid receptor antagonists. In 2021, the HISTOALDO consensus (histology of primary aldosteronism) and the routine use of immunohistochemistry (CYP11B2) made it possible to describe all the histopathological variations between a simple cortical adrenal tumour and bilateral hyperplasia.

Primary hyperaldosteronism due to unilateral or bilateral lesions with lateralised secretion (confirmed by venous sampling or NP53 scintigraphy) usually warrants surgical management via adrenalectomy.

However, while the effectiveness of the treatment is almost guaranteed to cure hypokalaemia, blood pressure changes after surgery remain highly variable, with few criteria available to predict the impact of surgery on blood pressure. Some patients are completely cured and can discontinue all antihypertensive medications, while others experience improvement, allowing a reduction in treatment. A final group shows no change in blood pressure post-adrenalectomy.

The main objective of this study is to evaluate the predictive value of measuring hormone status (aldosterone, renin and ARR) on the first day after surgery for postoperative blood pressure outcomes (clinical criteria: Systolic Blood Pressure).

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent unilateral adrenalectomy for primary hyperaldosteronism between 2017 and 2025.

Exclusion Criteria:

-none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent unilateral adrenalectomy for primary hyperaldosteronism between 2017 and 2025.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the predictive value of the evolution of the ARR between the preoperative period and Day 1 post-surgery on clinical blood pressure outcome | 2-3 months
  To evaluate the the evolution of the ARR between the preoperative period and Day 1 post-surgery predicts the clinical blood pressure outcome (clinical PASO criteria) observed two months after unilateral adrenalectomy for lateralized primary hyperald

SECONDARY OUTCOMES:
To evaluate the predictive value of ARR on Day 1 following unilateral adrenalectomy for primary hyperaldosteronism on clinical blood pressure outcome (clinical PASO criteria) | 2-3 months
To evaluate the predictive value of aldosterone levels on Day 1 following unilateral adrenalectomy for primary hyperaldosteronism on clinical blood pressure outcome (clinical PASO criteria) | 2-3 months
To evaluate the predictive value of renin levels on Day 1 following unilateral adrenalectomy for primary hyperaldosteronism on clinical blood pressure outcome (clinical PASO criteria) | 2-3 months
To determine whether intraoperative blood pressure variations during unilateral adrenalectomy for primary hyperaldosteronism predict postoperative clinical blood pressure outcome (clinical PASO criteria) | 2-3 months
To identify patient-related factors associated with postoperative clinical blood pressure outcome (clinical PASO criteria) | 2-3 months
To identify histopathological factors associated with postoperative clinical blood pressure outcome (clinical PASO criteria) | 2-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRERD, Study Director — CIC-P; Claire NOMINE-CRIQUI, PH, Principal Investigator — CVMC; Laurent BRUNAUD, PU-PH, Principal Investigator — CVMC

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vignaud T, Baud G, Nomine-Criqui C, Donatini G, Santucci N, Hamy A, Lifante JC, Maillard L, Mathonnet M, Chereau N, Pattou F, Caiazzo R, Tresallet C, Kuczma P, Menegaux F, Drui D, Gaujoux S, Brunaud L, Mirallie E; Eurocrine Study Group. Surgery for Primary Aldosteronism in France From 2010 to 2020 - Results from the French-Speaking Association of Endocrine Surgery (AFCE): Eurocrine Study Group. Ann Surg. 2023 Nov 1;278(5):717-724. doi: 10.1097/SLA.0000000000006026. Epub 2023 Jul 21. PMID 37477017
- [Background] Mete O, Erickson LA, Juhlin CC, de Krijger RR, Sasano H, Volante M, Papotti MG. Overview of the 2022 WHO Classification of Adrenal Cortical Tumors. Endocr Pathol. 2022 Mar;33(1):155-196. doi: 10.1007/s12022-022-09710-8. Epub 2022 Mar 14. PMID 35288842
- [Background] Amar L, Baguet JP, Bardet S, Chaffanjon P, Chamontin B, Douillard C, Durieux P, Girerd X, Gosse P, Hernigou A, Herpin D, Houillier P, Jeunemaitre X, Joffre F, Kraimps JL, Lefebvre H, Menegaux F, Mounier-Vehier C, Nussberger J, Pagny JY, Pechere A, Plouin PF, Reznik Y, Steichen O, Tabarin A, Zennaro MC, Zinzindohoue F, Chabre O. SFE/SFHTA/AFCE primary aldosteronism consensus: Introduction and handbook. Ann Endocrinol (Paris). 2016 Jul;77(3):179-86. doi: 10.1016/j.ando.2016.05.001. Epub 2016 Jun 15. PMID 27315757
- [Background] Williams TA, Lenders JWM, Mulatero P, Burrello J, Rottenkolber M, Adolf C, Satoh F, Amar L, Quinkler M, Deinum J, Beuschlein F, Kitamoto KK, Pham U, Morimoto R, Umakoshi H, Prejbisz A, Kocjan T, Naruse M, Stowasser M, Nishikawa T, Young WF Jr, Gomez-Sanchez CE, Funder JW, Reincke M; Primary Aldosteronism Surgery Outcome (PASO) investigators. Outcomes after adrenalectomy for unilateral primary aldosteronism: an international consensus on outcome measures and analysis of remission rates in an international cohort. Lancet Diabetes Endocrinol. 2017 Sep;5(9):689-699. doi: 10.1016/S2213-8587(17)30135-3. Epub 2017 May 30. PMID 28576687